CLINICAL TRIAL: NCT02482727
Title: BFR DISTRAD: Blood Flow Restricted Training During Rehabilitation Following Distal Radius Fracture Repair
Acronym: BFR DISTRAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jill Cancio, Jill Cancio, OTD, OTR, CHT, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C.2015.104
Record Dates: First submitted 2015-06-22; First posted 2015-06-26 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2016-07

CONDITIONS: Distal Radius Fracture; Rehabilitation
Keywords: Blood Flow Restriction; Occlusion training; Distal radius fracture
MeSH Terms: conditions — Wrist Fractures | interventions — Tourniquets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- non-occlusion training group (No Intervention): The control (non-occlusion training) group will follow the standard post-operative distal radius fracture rehabilitation protocol. Treatment will include passive, active assistive,active range of motion (P/AA/AROM) to wrist, forearm and hand; desensitization as needed; edema control as needed; heat/cold modalities as needed; and strengthening exercises.
- occlusion training with DELFI PTS ii tourniquet (Experimental): The occlusion training group will follow the same protocol as described above but will utilize occlusion training with the strengthening exercises. Investigators will use an established occlusion training protocol already being. Intervention: occlusion training with tourniquet (DELFI PTS ii portable tourniquet system)
  Interventions: Device: occlusion training with tourniquet (DELFI PTS ii portable tourniquet system)

INTERVENTIONS:
Device: occlusion training with tourniquet (DELFI PTS ii portable tourniquet system) — A cuff will be wrapped around the most proximal portion of the arm of the involved extremity. In order to individualize the pressure for each subject, the limb occlusion pressure will be measured (with dopplar ultrasound over the radial artery at the wrist level) at the first scheduled therapy visit. The cuff pressure utilized during the post-operative exercises will be set at 50% of the limb occlusion pressure. The subjects' strength will be re-assessed approximately every 2-4 weeks and the load will be increased as tolerated.
  Arms: occlusion training with DELFI PTS ii tourniquet

SUMMARY:
Occlusion training, resistance exercise performed with a specialized venous tourniquet, leads to beneficial changes in muscle strength at low resistance and minimal stress on the nearby joint. This novel resistance training has the potential to greatly improve muscle strength gains in individuals who are unable, for medical reasons, to perform the high resistance exercises typically required to improve strength. Our study will examine the effect of this technique on strength recovery following distal radius fracture repair. The primary objective of the intervention is to achieve accelerated recovery of forearm, wrist and hand function as assessed using measures such as grip/pinch strength, validated questionnaires, and functional outcome testing. Occlusion training can potentially serve as a specialty intervention for rehabilitation patients, reduce the cost of care, and improve the treatment options for both patients and providers.

DETAILED DESCRIPTION:
Investigators will perform a prospective, randomized, controlled study. All subjects in this group will be adults having undergone an open reduction internal fixation of the distal radius at San Antonio Military Medical Center (SAMMC) clinic system. Participants will be provided information about the study and inclusion/exclusion criteria, and upon conclusion of the formal consenting process, and signature of the consent document, will be considered enrolled in the study. Prior to initiation of any study procedures each patient must be cleared for participation in treatment by his or her surgeon as per standard post-operative protocol. This will be verified by accessing the medical record to confirm that a referral was made for post-operative rehabilitation. Before initiation of treatment, the enrolled subjects will be randomized to either a standard rehabilitation group or an occlusion training rehabilitation group. Treatment will be initiated approximately 6 weeks after surgery (when cleared by the orthopedic surgeon). Participants will undergo approximately 8-12 weeks of treatment with therapy sessions two to three days a week (consistent with standard of care), and will have re-assessments completed at approximately 4 weeks, 8 weeks, and 12 weeks after initiating the training protocol. The 12-week time point (after initiation of therapy) will be at approximately the same time that patients are released for full activity per standard of care.

The control (non-occlusion training) group will follow the standard post-operative distal radius fracture rehabilitation protocol. Treatment will include passive, active assistive, active range of motion (P/AA/AROM) to wrist, forearm and hand; desensitization as needed; edema control as needed; heat/cold modalities as needed; and strengthening exercises. Specific strengthening exercises which include wrist flexion/extension over a foam wedge, forearm pronation/supination with arm positioned at side and elbow at 90 degrees, thumb opposition as well as grip strengthening.

The occlusion training group will follow the same protocol as described above but will utilize occlusion training with the strengthening exercises. Investigators will use an established occlusion training protocol already being used at the CFI. The resistance for strength training will be determined based on the individual participants tolerance.. A cuff will be wrapped around the most proximal portion of the arm of the involved extremity. In order to individualize the pressure for each subject, the limb occlusion pressure will be measured (with dopplar ultrasound over the radial artery at the wrist level) at the first scheduled therapy visit. The cuff pressure utilized during the post-operative exercises will be set at 50% of the limb occlusion pressure. Repetitions will be 30, 15, 15 and 15 for each of the four sets. A 30-second rest will be given between sets. The tourniquet will stay inflated throughout the entire exercise and rest sessions, and no longer than 30 minutes consecutively for any time that the tourniquet is inflated. After completion of the 4 sets the tourniquet pressure will be deflated. The subjects' strength will be re-assessed approximately every 2-4 weeks and the load will be increased as tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Status post open reduction internal fixation for a distal radius fracture
* Males and females 18-65 years of age
* Eligible to receive care at Military Treatment Facilities (DEERS eligible)
* Must be able to read and write in English in order to consent

Exclusion Criteria:

* Contralateral upper extremity involvement resulting in less than normal range of motion, muscle strength, or daily pain greater than 1/10.
* Pregnancy - per patient self-report. Due the expected small number of pregnant individuals and resulting inability to account for its effect on resulting outcomes, these patients will not be included in the study.
* Recent history of deep vein thrombosis, within the 12 months or on active treatment with anticoagulants
* History of upper quadrant lymph node dissection
* History of endothelial dysfunction
* Patient endorsement of easy bruising
* Active Infection
* Cancer (current diagnosis per medical record)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Grip strength | 18 weeks
  grip strength measured with the JAMAR Hand Dynamometer. The mean of three successive trials will be recorded

SECONDARY OUTCOMES:
Pinch strength | 18 weeks
  Pinch strength will be assessed using the PG-60 Pinch Gauge.The mean of three successive trials will be recorded for each pinch position (tip, key and palmar)
Joint range of motion | 18 weeks
  Joint range of motion (ROM) will be assessed using a plastic goniometer, an inexpensive device with two plastic arms that are aligned with relevant body segments to provide joint angle information. Forearm, wrist radial/ulnar deviation and hand ROM will be assessed according to the guidelines recommended by the American Society for Hand Therapy

OTHER OUTCOMES:
Performance measure DASH | 18 weeks
  The Disabilities of the Arm, Shoulder and Hand (DASH) )is a 30-item self-report measure that assesses a subject's perceived ability to complete twenty-one upper extremity functional activities using a 5-point Likert scale. The cumulative DASH score is scaled from 0 to 100, with higher scores indicating increased disability
Performance measure PRWE | 18 weeks
  The Patient Rated Wrist Evaluation (PRWE) is a 15-item questionnaire that assesses wrist pain (5 items) and disability (10 items) in activities of daily living
Performance measure JTHFT | 18 weeks
  The Jebsen-Taylor Hand Function Test (JTHFT) is a seven part test that evaluations the time needed to perform seven hand-related tasks
Performance measure PSFS | 18 week
  The Patient Specific Functional Scale (PSFS) is a patient-specific outcome measure to assess functional status[52]. The patient is asked to identify three to five activities that he or she has difficulty performing due to his or her condition. The patient then rates the amount of limitation he or she has in performing each of these activities on an 11-point scale with 0 being unable to perform the activity and 10 being able to perform the activity with no problem. An average score for the activities gives an ability score out of 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States